CLINICAL TRIAL: NCT04453215
Title: The Effect of Dental Laser Therapy for Patients With Systemic Lupus Erythematosus
Brief Title: Laser Therapy for Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Merve Benli (Other)
Responsible Party: Sponsor-Investigator, Dr. Merve Benli, Assistant Professor, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1298
Record Dates: First submitted 2020-06-28; First posted 2020-07-01 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Systemic Lupus Erythematosus; Muscle Pain; Chewing Function
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myalgia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- test group (Experimental): SLE patients treated with infrared laser irradiation
  Interventions: Device: GaAlAs semiconductor diode laser device
- placebo group (Placebo Comparator): SLE patients treated with red laser irradiation
  Interventions: Device: GaAlAs semiconductor diode laser device
- control group (No Intervention): no therapy group

INTERVENTIONS:
Device: GaAlAs semiconductor diode laser device — low-level laser therapy
  Arms: placebo group; test group

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic, autoimmune disease that has detrimental effects on connective tissue and other organs. The musculoskeletal system is one of the most affected systems in this group of patients including the temporomandibular joint. The most common symptoms when muscle involvement in SLE are muscle atrophy decreased muscle strength and myopathy. SLE activity and long-term corticosteroid use are thought to be responsible for these symptoms, thus, SLE patients are accepted to be at higher risk for temporomandibular joint disorders (TMD). Low-level laser therapy(LLLT) is frequently used in the treatment of TMD due to its pain relief and anti-inflammatory effect. Thus, in this study, LLLT has been used to evaluate this treatment modality on the chewing function and pain values of SLE patients with myogenic TMD.

ELIGIBILITY:
Inclusion Criteria:

* Having myogenic temporomandibular joint disorder,
* Following a stable medical regime,
* Showing minimum pain intensity of 50 mm on the visual analog scale.

Exclusion Criteria:

* Having concurrent systemic diseases,
* Using antimalarial drugs,
* Wearing removable prosthesis,
* History of facial trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
pain value | 2 months
  Pain intensity was evaluated by using Visual Analog Scale(VAS).
chewing function | 2 months
  The chewing function was evaluated by measuring the geometric mean diameter of crushed test food.

CONTACTS AND LOCATIONS:
Overall Officials: merve benli, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Istanbul university,Faculty of Dentistry, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When requested by a researcher, the data can be shared without the identity of the patient.
Supporting Information: Study Protocol
Time Frame: The data will become available when confirmed, and it will be available for one year.
Access Criteria: The study protocol and patient selection will be shared.